CLINICAL TRIAL: NCT06536517
Title: A Randomized Controlled Trial to Study the Effects of One-time Intra-operative Dosing of Methadone During Laparoscopic or Robotic Hysterectomy in Reducing Opioid Prescription.
Brief Title: The Effects of One-time Intraoperative Methadone During Laparoscopic Hysterectomy in Reducing Opioid Prescription.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00459067
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Fibroid Uterus
Keywords: hysterectomy; methadone; opioids
MeSH Terms: conditions — Leiomyoma | interventions — Methadone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methadone (Experimental): Intra-operative single dose IV Methadone (0.25 mg/kg of ideal body weight)
  Interventions: Drug: Methadone
- Short-Acting Opioid (Other): Standard intra-operative IV shorter acting opioids
  Interventions: Drug: Methadone

INTERVENTIONS:
Drug: Methadone — Intra-operative single dose IV Methadone (0.25 mg/kg of ideal body weight)

SUMMARY:
Currently, there is a nationwide epidemic of opioid abuse and overdose deaths. One source of excess opioids is overprescribing in the postoperative period. This study aims to find the optimal pain medication plan during and after laparoscopic hysterectomy to eliminate long-term opioid use.

Given the increasing opioid abuse and over-prescription post-operatively, an effort should be made to determine whether one time dosing of Methadone, a longer opioid analgesics, intra-operatively is an adequate potential in treating postoperative pain after hysterectomy surgeries. The investigators hypothesize that this could minimize the need for additional post-operative and outpatient opioid prescriptions and decrease the adverse effects that are associated with the consumption, including new opioid abuse.

Intervention group will receive methadone intraoperatively while the other group would receive short-acting opioids (standard).

DETAILED DESCRIPTION:
Problem:

The relief of moderate to severe postoperative pain in surgeries including abdominal surgeries continues to pose a major therapeutic dilemma. The traditional and most common therapy is the administration of short-acting opioid analgesics, intra-operative and post-operative, at intervals every 3-4 hours. However, the use of opioids with relatively short plasma half-lives at varying intervals may lead to various fluctuating drug concentrations in plasma, and side effects including respiratory, longer hospitalizations, delayed ambulation, inadequate pain relief and potential avenues for abuse. Identifying a more efficient and safer therapy for intraoperative pain analgesia can be helpful in controlling pain requirements in the post-operative setting.

In major inpatient and ambulatory surgeries, intraoperative single-dose methadone, through its unique pharmacology, has been shown to produce better analgesia, reduce opioid use and minimize adverse side effects compared with conventional repeated dosing of short-duration opioids. Additionally, methadone is theorized to be an N-methyl-D-aspartate (NMDA) receptor noncompetitive antagonist, which may contribute to its increase in analgesic potential as compared with fentanyl analogues. Finally, it has been shown to improve ambulation in the post operative anesthesia setting and pain control in chronic pain patients. The study of intra-operative methadone has not been extensively studied for gynecology surgeries, but one study has shown the decrease of mean opioid consumption post operatively after receiving one dose of intra-operative methadone compared to shorter acting opioids in same-day laparoscopic myomectomy. Given the increasing opioid abuse and over-prescription post-operatively, an effort should be made to determine whether one time dosing of longer opioid analgesics intra-operatively is an adequate potential in treating postoperative pain after hysterectomy surgeries and could minimize the need for additional post-operative and outpatient opioid prescriptions.

This study aims at addressing the requirement for postoperative opioid prescription after intraoperative longer acting vs shorter acting opioids in laparoscopic hysterectomy.

Hypothesis:

Single dose of intra-operative methadone is an adequate potential in treating post-operative pain after laparoscopic total hysterectomy surgeries, reducing the additional need for post-operative and outpatient opioid prescriptions and decreasing the adverse effects associated with opioid consumption.

Importance of research:

Given the increasing opioid abuse and over-prescription post-operatively, an effort must be made to determine whether one time dosing of longer opioid analgesics intraoperatively in conjunction with non-opioid multimodal medications is adequate to treat postoperative pain after laparoscopic hysterectomy. Additionally, this intervention may decrease the need for additional prescriptions or unscheduled patient contacts.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a uterus
* Age 18 years old and above
* Undergoing minimally invasive (laparoscopic or robotic) hysterectomy with ovarian preservation
* Benign indications for hysterectomy
* Agreeing to participate

Exclusion Criteria:

* Chronic pain syndromes patients including fibromyalgia
* Patients currently on long-term (i.e. for more than three months) opioid use
* Patients currently on agonist-antagonist medications (e.g. buprenorphine)
* Patients taking a selective serotonin reuptake inhibitor or monoamine oxidase inhibitor
* Conversion to laparotomy
* Allergy or other contraindication to the prescribed medications such as methadone, fentanyl, acetaminophen or oxycodone
* Severe Obstructive Sleep Apnea (OSA)
* Pregnant/breastfeeding patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Total post-operative opioid requirements in oral morphine milligram equivalents (MME) | 1 week
  Total post-operative opioid requirements in oral morphine milligram equivalents (MME) in first 7 post operative days.

SECONDARY OUTCOMES:
Mobility and satisfaction of analgesia | Post operative day 1, Post operative day 7
  Mobility and satisfaction of analgesia on post-operative day one and seven (binary question Y/N)
Number of unplanned returns to emergency room/clinic or patient initiated phone call regarding pain | 1 week
Overall satisfaction with pain control | 1 week
  0-10 scale (0- no pain, 10-worst pain)

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Borahay, MD, MBA, PhD, Principal Investigator — Study Principal Investigator
Locations (2):
- United States (2):
  - The Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - The Johns Hopkins Hospital, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No